CLINICAL TRIAL: NCT03705364
Title: Validation of a Fall Prevention Program Among Non-Ambulatory Wheeled Mobility Device Users With Multiple Sclerosis
Brief Title: Fall Prevention Program for Non-ambulatory Wheeled Mobility Device Users Living With MS
Acronym: iRoll
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18124
Record Dates: First submitted 2018-02-27; First posted 2018-10-15 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
Keywords: wheelchair; non-ambulatory
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait List Control Group (No Intervention): Wait list control group
- Fall Management program (Experimental): Intervention arm
  Interventions: Other: Fall Management program

INTERVENTIONS:
Other: Fall Management program — Comprehensive fall management program that develops strategies for non-ambulatory wheelchair users living with MS to develpo strategies to recover from a fall.
  Arms: Fall Management program

SUMMARY:
A research study to examine the effectiveness of a fall management program to prevent falls and develop fall recovery strategies for wheeled mobility device users living with Multiple Sclerosis.

DETAILED DESCRIPTION:
Falls are a serious concern for wheelchair and scooter users with Multiple Sclerosis (MS). Approximately 75% of the population reports at least one fall in a 6-month period and nearly half report frequent falls. Falls can result in physical injuries and contribute to activity curtailment. Despite the negative consequences, limited evidenced-based fall prevention programs designed specifically for wheelchair and scooter users with MS exist.

Recognizing the threat falls pose to health and well-being and the dearth of fall prevention programs, the purpose of this study to perform a structured process evaluation and examine the feasibility and efficacy of a community-based intervention specifically designed to reduce fall incidence among wheelchair and scooter users with MS. Secondary aims of the intervention are to improve functional mobility skills associated with fall risk (e.g. transfer and wheelchair skills, balance), increase knowledge of fall risk factors, decrease fear of falling and enhance quality of life and community participation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Multiple Sclerosis
2. >18 years old
3. Main form of mobility is via a wheeled mobility device (Patient Determined Disease Steps Level 7)
4. Self reported ability to transfer with moderate assistance or less
5. Self-reported fall history (at least 1 fall/12 months)

Exclusion Criteria:

1. MS exacerbation in the past 30 days
2. Received a score of 10 or above to the Short Blessed Test (attached)
3. Inability to sit upright for at least 1 hour.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in fall incidence | 44 weeks
  Fall Diary; Construct: to report and track the number of falls experienced; Less number of falls indicates better outcome.

SECONDARY OUTCOMES:
Management of Fall | 44 weeks
  Fall Management Scale (FMS); Construct: to measure the perceived ability to manage risk of falls or actual falls; Scale range: 5 - 45, higher scores indicate lower degree of confidence; Items are summed to get the final score.
Prevention of Fall | 44 weeks
  Falls Prevention Strategies Survey (FPSS); Construct: to measure the use of fall prevention strategies; Scale range: 0 - 22, higher scores reflect more regular use of more fall prevention strategies; Never do: 0, Do sometimes: 1, Do regularly: 2; Items are summed to get the final score.
Prevention and Management of Fall | 44 weeks
  Falls Prevention and Management Questionnaire (FPMQ); Construct: to measure the ability to prevent and manage falls; Scale range: 0 - 48, higher scores indicate higher ability to prevent and manage falls; Items are scored from 0 ("strongly disagree") to 4 ("strongly agree"); Items are summed to get the final score.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Rice, PhD,MPT,ATP, Principal Investigator — Department of Kinesiology and Community Health, College of Applied Health Sciences, University of Illinois at Urbana-Champaign
Locations (3):
- United States (3):
  - The Shepherd Center, Atlanta, Georgia
  - UIC, Chicago, Illinois
  - UIUC, Urbana, Illinois

IPD SHARING:
Plan to Share IPD: No
Individuals participant data will not be available to other researchers.

REFERENCES:
- [Derived] Rice LA, Peterson EW, Backus D, Sung J, Yarnot R, Abou L, Van Denend T, Shen S, Sosnoff JJ. Validation of an individualized reduction of falls intervention program among wheelchair and scooter users with multiple sclerosis. Medicine (Baltimore). 2019 May;98(19):e15418. doi: 10.1097/MD.0000000000015418. PMID 31083170

DOCUMENTS (1):
  • Informed Consent Form (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT03705364/ICF_000.pdf